CLINICAL TRIAL: NCT06666361
Title: Health Literacy and Health Promotion Behaviors Among Middle-aged and Older Adults with Hypertension in Rural Communities: a Mixed Methods Study
Brief Title: Middle-aged and Older Adults with Hypertension in Rural Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, HSIAO,SU-CHIU, Chi Mei Medical Center,Liouying, Director Nursing Department, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMMC11309-L01; IRB Serial No.: 11309-L01 (Registry Identifier: ChiMei Institutional Review Board)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
Keywords: Hypertension; rural; health literacy; health promotion; middle-aged and older adults
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group:receiving intervention (Experimental): The experimental group participates in the Mobio Health Multimedia Hypertension Education Program, which includes a hypertension health education manual and a mobile health (m-health) intervention, aimed at enhancing participants' health literacy and promoting health-enhancing behaviors.
  Interventions: Other: Experimental Group
- Control group :Non intervention (Experimental): In the control group, participants received the same hypertension health education manual as the experimental group.
  Interventions: Other: control group

INTERVENTIONS:
Other: Experimental Group — The experimental group participates in the Mobio Health Multimedia Hypertension Promotion Program, which includes a hypertension education manual and a mobile health (m-health) intervention aimed at enhancing participants' health literacy and promoting healthy behaviors. In the first week, participants receive the health-education manual on-site, with face-to-face explanations and guidance on using mobile resources, such as text messaging, provided by the Sub-Investigator.
  The mobile health intervention transforms the manual's content into six video units, each covering a specific topic, and these videos are continuously pushed over a two-month period. Distributed through LINE@, the official LINE account of the nursing platform, participants can easily access information via the chat menu at the bottom of the screen. This setup improves accessibility, making it convenient for participants to locate and use essential health information directly from the chat window.
  Arms: Experimental Group:receiving intervention
Other: control group — The control group received one copy of the same health education manual as the experimental group. The sub-Investigator only explained how to use the manual, and afterwards, no face-to-face teaching or m-Health interventions were conducted. After the experiment concluded, the m-Health program used by the experimental group would be provided to the control group.
  Arms: Control group :Non intervention

SUMMARY:
Does the m-Health intervention have a positive effect on the health literacy and health promotion behaviors of the study participants?

DETAILED DESCRIPTION:
This study adopted a mixed methods study, and the first stage was a qualitative research design. The second phase was a quantitative research design aims to evaluate the effectiveness of applying healthy lifestyle intervention on the health literacy and health promotion behaviors among middle-aged and older adults with hypertension in rural communities. Recruitment is planned to be conducted in the cardiology outpatient clinic of a regional teaching hospital in the south. It will be a random assignment, single-blind, experimental research design, using simple random sampling to assign to the experimental group and the control group (experimental group: hypertension health education manual + m-Health; control group: hypertension health education manual), a two- month intervention program was carried out, and the questionnaire survey was conducted three times: once as a pre-test and twice as post-tests (during the 4th week and the 8th week of the intervention). Data analysis was conducted using statistical software (SPSS, version 22.0) for data management and statistical analysis, and analysis was conducted using descriptive statistics, independent sample t-test, chi-square test, and generalized estimating equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hypertension for one year or more (including) and controlled with medication (systolic blood pressure ≥ 130 mmHg and diastolic blood pressure ≥ 80 mmHg).
2. Aware hypertensive patients aged ≥ 45 years with the ability to read and write.
3. Able to take medication independently.
4. Own a smartphone and are able to use it, and are willing to receive text messages (TxtM) or mobile health interventions (m-Health).
5. Agree to participate in the study.

Exclusion Criteria:

1. Have cognitive impairments or mental disorders.
2. CCI (Charlson Comorbidity Index) score ≥ 3.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1.To explore the effectiveness of mobile health(m-health) interventions on the health literacy of study participants. 2.To explore the effectiveness of mobile health(m-health) interventions on the health promotion behaviors of study participants. | 1.Total duration for Each Participant: 2 months Intervention Period: From December 2024 to December 2025
  A structured questionnaire survery was administered at the start, and at the 4th and 8th weeks of the intervention to evaluate its effectiveness. The questionnaire includes:(1) The Hypertension Health Literacy Scale, with scores ranging from 10 to 40, where higher scores indicate better outcomes; (2) The short-form Chinese Health-Promoting Lifestyle Profile, with scores ranging from 24 to 96, where higher scores indicate better outcomes.

SECONDARY OUTCOMES:
1.To explore the factors influencing the health literacy of study participants. 2.To explore the factors influencing the health promotion behaviors of study participants. | 1.Total duration for Each Participant: 2 months Intervention. 2.Period: From December 2024 to December 2025
  A structured questionnaire was administered at the start, at weeks 4 and 8 of the intervention, and for post-intervention evaluation. The details are as follows: (1) Basic Characteristics, including age , gender, height (cm), weight (kg), BMI(weight and height will be combined to report BMI in in kg/m²), education, marital status, residential area, employment, economic status, living situation, clinic transportation, duration of hypertension, regular medication, and presence of other chronic diseases; (2) Hypertension Knowledge Scale( 0 to 10, higher scores = greater knowledge); (3) Adherence to Refills and Medications Scale (12-48, higher scores = better outcomes); (4) System Usability Scale, graded as: A (90-100), B (80-89), C (70-79), D (60-69), and F (0-59), with strong face validity and an average score of about 70; scores above 70 are considered acceptable; (5) Learning Satisfaction Questionnaire (12-60, higher scores= better outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Su.Chiu Hsiao, Principal Investigator — Chi Mei Medical Center,Liouying Director Nursing Department
Locations (1):
- Chi Mei Hospital, Liouying, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No